CLINICAL TRIAL: NCT01217450
Title: A Phase 1 Study of AZD6244 in Combination With Cetuximab in Refractory Solid Tumors
Brief Title: Selumetinib and Cetuximab in Treating Patients With Refractory Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02915; NCI-2012-02915 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000686619; CO10901 (Other: University of Wisconsin Medical School); 8627 (Other: CTEP); P30CA014520 (NIH); U01CA062491 (NIH)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2013-12

CONDITIONS: Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — AZD 6244; Cetuximab

ARMS (1):
- Treatment (selumetinib, cetuximab) (Experimental): Patients receive oral MEK inhibitor AZD6244 once or twice daily on days 1-28 and cetuximab IV over 60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: selumetinib; Biological: cetuximab; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: selumetinib — Given orally
  Other Names: ARRY-142886; AZD6244
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and the best dose of MEK Inhibitor AZD6244 when given together with cetuximab in patients with advanced or refractory solid tumors that cannot be removed by surgery. MEK inhibitor AZD6244 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving MEK Inhibitor AZD6244 together with cetuximab may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the dose limiting toxicities and the maximum tolerated dose of AZD6244 in combination with cetuximab in advanced, refractory solid tumors.

II. To assess for evidence of anti-tumor activity with this combination, per tumor measurements using RECIST criteria.

SECONDARY OBJECTIVES:

I. To evaluate the pharmacokinetics of AZD6244 and cetuximab when administered concomitantly.

II. To evaluate the safety and tolerability of the combination of AZD6244 and cetuximab in patients with K-RAS mutated metastatic colorectal cancer.

TERTIARY OBJECTIVES:

I. To assess the inhibition of the RAF/MEK/ERK pathway in peripheral blood mononuclear cells secondary to treatment with AZD6244.

II. To evaluate the pharmacokinetics of AZD6244 in combination with cetuximab and the relation to treatment side effects.

OUTLINE: This is a dose-escalation study of MEK inhibitor AZD6244.

Patients receive oral MEK inhibitor AZD6244 once or twice daily on days 1-28 and cetuximab IV over 60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and periodically during study for pharmacokinetic and biomarker analyses.

After completion of study treatment, patients are followed up for 1 month or every 3 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* In the dose escalation cohorts: Patients must have histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative measures do not exist or are no longer effective; histology can be based on either the primary tumor or metastases
* In the MTD expansion cohort: Patients must have biopsy proven K-RAS mutant, metastatic colorectal cancer that has progressed on at least 2 prior standard therapies; K-RAS mutation status must be verified by a CLIA-certified laboratory (NOTE: colorectal patients enrolled during the dose escalation portion do not need to be K-RAS mutant in order to be eligible)
* Patients must be at least 4 weeks since prior chemotherapy, 6 weeks if the last regimen included nitrosureas or mitomycin C; prior radiation is allowed as long as the radiation was completed 4 weeks prior to study treatment and no more than 35% of marrow irradiated
* ECOG performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal (AST and ALT =< 5.0 X institutional upper limit of normal will be permitted if liver metastases are present)
* Creatinine =< 1.5 X institution upper limit of normal OR creatinine clearance >= 45 mL/min/1.73 m^2, as calculated by Cockroft-Gault formula, for patients with creatinine levels above institutional normal
* Patients may have received prior cetuximab
* The effects of AZD6244 on the developing human fetus are unknown; for this reason and because small molecule kinase inhibitors as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception prior to study entry and for 16 weeks following the last dose of study treatment. Acceptable methods of birth control include implants, injectables, combined oral contraceptives, (which must all be combined with barrier methods of contraception), some IUDs, sexual abstinence, and vasectomized partner; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document
* Patients with brain metastases that have been treated and stable for 2 months will be eligible for this study
* Subjects undergoing anti-coagulation therapy with LMWH and warfarin are eligible; subjects receiving both warfarin and AZD6244 should have more frequent PT/INR monitoring

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy or hormonal therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered (=< grade 1) from adverse events due to agents administered more than 4 weeks earlier
* Concurrent treatment with an investigational agent other than the investigational agent(s) used in this study OR treatment within 4 weeks of study entry with any investigational agent(s) or device(s)
* Failure to recover fully (as judged by the investigator) from prior surgical procedures
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD6244 or other agents used in study
* Patients taking high doses (more than recommended daily dose) of vitamin E will be excluded; patients can discontinue use of high dose vitamin E prior to study entry to be considered eligible
* Any condition (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease) that impairs their ability to swallow and retain AZD6244 capsules
* Patients with malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel are excluded; subjects with ulcerative colitis, inflammatory bowel disease, or a partial or complete small bowel obstruction are also excluded
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, prior cardiomyopathy, LVEF < 50%, unstable angina pectoris, cardiac arrhythmia (i.e. atrial fibrillation), or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because AZD6244 is a small molecule kinase inhibitor with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD6244, breastfeeding should be discontinued if the mother is treated with AZD6244; these potential risks may also apply to other agents used in this study
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD6244; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients who are serologically positive for Hepatitis B or C, or have a history of liver disease, other forms of hepatitis or cirrhosis are ineligible
* Use of strong CYP1A2 or 3A4 inducers and/or inhibitors (for example, but not limited to, ketoconazole, rifampicin, atazanavir, clarithromycin, indinavir, itraconazole, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, troleandomycin (TAO), voriconazole, grapefruit or grapefruit juice, rifabutin, rifapentine, phenytoin, carbamazepine, phenobarbital and St. John's Wort) is not permitted while on study or within 7 days prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
MTD of selumetinib combined with cetuximab | 28 days
  Graded using the NCI Common Toxicity Criteria.
Tumor response, as evaluated by the RECIST | Up to 4 weeks after completion of study treatment
  Analyzed by descriptive statistics, and summarized in tabular format. 95% confidence intervals will be computed using the method proposed by Chang.

SECONDARY OUTCOMES:
Toxicities graded using the NCI Common Toxicity Criteria | Up to 4 weeks after completion of study treatment
  Summarized in terms of types and severities. Analyzed descriptively in tabular format. Ninety percent confidence intervals for the proportions of patients with complications (grade 3 or higher toxicities) will be constructed using the Wilson's score method.

CONTACTS AND LOCATIONS:
Overall Officials: William Schelman, Principal Investigator — University of Wisconsin Medical School
Locations (3):
- United States (3):
  - National Cancer Institute Medicine Branch, Bethesda, Maryland
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Wisconsin Clinical Cancer Center, Milwaukee, Wisconsin